CLINICAL TRIAL: NCT04827641
Title: Severity Grading of Unexpected Events in Pediatric Surgery - Evaluation of Five Classification Systems and the Comprehensive Complication Index (CCI®)
Brief Title: Severity Grading of Unexpected Events in Pediatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Omid Madadi-Sanjani, Dr., Consultant, Center of Pediatric Surgery, Hannover Medical School
Other Study IDs: 2739-2015
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Complication of Surgical Procedure
Keywords: complications; unexpected events; severity grading systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Severity Grading assessment in children with perioperative unexpected events — Systematic documentation of all unexpected events was carried out by designated team members during daily routine team conferences. Briefly, on-call team members and all other staff reported on any unexpected event that had occurred within the previous 24 hours, after weekends during the past 72 hours. Events included those that had occurred in inpatients, outpatients and in the pediatric emergency department. Data concerning each event included patient demographics, diagnoses, treatments/operations and types of events.
  Other Names: According to Clavien-Dindo Classification; According to T92 Classification; According to contracted Accordion Classification; According to extended Accordion Classification; According to MSKCC Classification; According to Comprehensive Complication Index (CCI®)

SUMMARY:
Data on all patients who experienced unexpected events at the Department of Pediatric Surgery Hannover Medical School from 1st January 2017 to 30th November 2020 were documented prospectively. The department represents the only tertiary academic institution of the german province of Lower-Saxony (8 million inhabitants). The clinical spectrum of the department includes surgery of the neonate, gastrointestinal, hepatobiliary, thoracic and oncological surgery and pediatric urology.

ELIGIBILITY:
Inclusion Criteria:

* All patients with unexpected events during the in-hospital stay, in outpatient clinics and in the pediatric emergency department
* Informed consent was obtained from the legal guardian´s at admission

Exclusion Criteria:

* If no informed consent was obtained from the legal guardian´s at admission

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Data on all patients (preterm infants to 18 years of age) who experienced unexpected events at the Department of Pediatric Surgery Hannover Medical School from 1st January 2017 to 30th November 2020 were documented prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through study completion, an average of 3 years
  All adverse events were prospectively documented

SECONDARY OUTCOMES:
Categorization of adverse events | Through study completion, an average of 3 years
  Events associated with surgical/non-surgical interventions and events not associated with interventions such as organizational problems, management problems or underlying disease were differentiated.
Classification of adverse events | Through study completion, an average of 3 years
  According to the Clavien-Dindo-, T92-, contracted Accordion-, Extended Accordion- and MSKCC-Classification
Calculation of the Comprehensive Complication Index (CCI®) | 3 months
  Using an online tool based on the protocol by Staiger et al.(http://www.cci.assessurgery.com).

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sethi MV, Zimmer J, Ure B, Lacher M. Prospective assessment of complications on a daily basis is essential to determine morbidity and mortality in routine pediatric surgery. J Pediatr Surg. 2016 Apr;51(4):630-3. doi: 10.1016/j.jpedsurg.2015.10.052. Epub 2015 Oct 27. PMID 26628204
- [Background] Staiger RD, Cimino M, Javed A, Biondo S, Fondevila C, Perinel J, Aragao AC, Torzilli G, Wolfgang C, Adham M, Pinto-Marques H, Dutkowski P, Puhan MA, Clavien PA. The Comprehensive Complication Index (CCI(R)) is a Novel Cost Assessment Tool for Surgical Procedures. Ann Surg. 2018 Nov;268(5):784-791. doi: 10.1097/SLA.0000000000002902. PMID 30272585
- [Background] Staiger RD, Gerns E, Castrejon Subira M, Domenghino A, Puhan MA, Clavien PA. Can Early Postoperative Complications Predict High Morbidity and Decrease Failure to Rescue Following Major Abdominal Surgery? Ann Surg. 2020 Nov;272(5):834-839. doi: 10.1097/SLA.0000000000004254. PMID 32925252
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Strasberg SM, Linehan DC, Hawkins WG. The accordion severity grading system of surgical complications. Ann Surg. 2009 Aug;250(2):177-86. doi: 10.1097/SLA.0b013e3181afde41. PMID 19638919
- [Result] Zoeller C, Kuebler JF, Ure BM, Brendel J. Incidence of complications, organizational problems, and errors: Unexpected events in 1605 patients. J Pediatr Surg. 2021 Oct;56(10):1723-1727. doi: 10.1016/j.jpedsurg.2020.12.004. Epub 2020 Dec 13. PMID 33353740